CLINICAL TRIAL: NCT02199470
Title: β-cell Function in Type Diabetes May Not Be As Low As Presumed
Brief Title: β-cell Function in Type 1 Diabetes May Not Be As Low As Presumed
Status: Completed | Type: Observational
Sponsor: Gonca Incemehmet Tamer (Other)
Responsible Party: Sponsor-Investigator, Gonca Incemehmet Tamer, Istanbul Medeniyet University, Goztepe Research and Training Hospital, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: MUGEAH-1
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: TYPE 1 DIABETES
Keywords: β-CELLS,; MIXED MEAL TEST,; C-PEPTİDE
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum c-peptide levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- C-peptide minimal detectable: C-peptide level between 0,01-0,08 ng/mL
- C-peptide sustained: C-peptide level between higher or equal to 0,08 ng/mL
- C-peptide not detectable: C- peptide level equal to or lower than 0,01 ng/mL

SUMMARY:
Enhancing endogenous insulin production in type 1 diabetic patients (T1DP) can improve glycemic control and decrease complications and rates of mortality. However, it can be succesfull even if sufficient β-cell function is present. We aimed to evaluate the extent of β-cell function by determining fasting levels of C-peptide and those after meal stimulus.

DETAILED DESCRIPTION:
Background and aims: Enhancing endogenous insulin production in type 1 diabetic patients (T1DP) can improve glycemic control and decrease complications and rates of mortality. However, it can be succesfull even if sufficient β-cell function is present. We aimed to evaluate the extent of β-cell function by determining fasting levels of C-peptide and those after meal stimulus.

Materials and Methods: One hundred and thiryfive T1DP were planned to enrolı to the study. Ethics comittee of our hospital approved the study protocol, which was in accordance with the Helsinki Declaration. Fasting C-peptide levels of all participants and stimulated (at 90 th minute post mixed meal) C-peptide levels of 54 will be measured by using an electrochemiluminescence assay. Two categorizations will be done using fasting (the first categorization ) and at 90th minute post mixed meal test (the second categorization) of C-peptide levels. For the first categorization; the groups will be classified as follows: patients with undetectable ≤0.1 ng/mL (group 1); with minimal 0.1-0.8 ng/ml (group 2); and with sustained ≥0.8 ng/mL(group 3) C-peptide levels. For the second categorization, groups will be as follows: patients with undetectable ≤0.1 ng/mL (group 1); with minimal 0.1-0.8 ng/ml (group 2); and with sustained ≥0.8 ng/mL (group 3) C-peptide levels which increased at the 90th minute after the meal ≥150% of fasting C-peptide level.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients who have accepted to have mixed meal tolarance test

Exclusion Criteria:

* Patients with type 2 diabetes,
* patients with MODY

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
We aimed to evaluate the extent of β-cell function by determining fasting levels of C-peptide and those after meal stimulus. | 1 day (the duration of mixed test is 90 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Incemehmet Tamer, I, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Medeniyet University Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Joslin Medalist Study — http://creativecommons.org/licenses/by-nc-nd/3.0/